CLINICAL TRIAL: NCT03655353
Title: A Multicenter Phase II/III-study of 68Ga-ABY-025 PET for Non-invasive Quantification of HER2-expression in Advanced Breast Cancer
Brief Title: A Study of 68Ga-ABY-025 PET for Non-invasive Quantification of HER2-expression in Advanced Breast Cancer
Acronym: Affibody-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henrik Lindman (Other)
Collaborators: Roche Pharma AG (Industry); Swedish Cancer Society (Other); Affibody (Industry); Swedish Breast Cancer Group (Other)
Responsible Party: Sponsor-Investigator, Henrik Lindman, Coordinating Investigator, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABY-025-MI301
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Masking Description: Investigators will determine HER2 expression by ABY-PET without knowledge of the results from the biopsies (in Phase III part).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABY-PET (Experimental): 68Ga-ABY-025 is used as tracer for PET scan
  Interventions: Diagnostic Test: ABY-PET

INTERVENTIONS:
Diagnostic Test: ABY-PET — Diagnostic PET for HER2 expression

SUMMARY:
A large multi- center phase II/III study with 68Ga-ABY-025 PET and biopsies in patients with advanced HER2-positive breast cancer, where the primary endpoint of the study is to find out the correlation between the HER2 expression measured by 68Ga-ABY-025 PET and standard histopathology from relevant tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age ≥18 years.
3. Histologically or cytologically confirmed HER2-positive or borderline positive (for definition see below) adenocarcinoma of the breast.

   HER2-positive defined as:
   1. 3+ by immunohistochemistry [IHC] in >10% of cell areas.
   2. 2+ by IHC in >10% of cell areas and HER2/CEP17 ratio ≥2.0 or HER2 copy number ≥ 6.0 by in situ hybridization [ISH]).

      HER2-borderline positive defines as:
   3. 2+ by IHC and HER2/CEP17 ratio <2.0 and/or HER2 copy number 4.0 - 6.0 by in situ hybridization [ISH]) ("equivocal").
   4. 2+ by IHC and HER2/CEP17 ratio <2.0 and/or HER2 copy number <4.0 by in situ hybridization [ISH]) ("2+ ISH negative").
   5. Known inhomogeneous HER2-expression in the primary tumor with HER2-positive areas <10% ("inhomogeneous").
4. Primary breast cancer planned for neoadjuvant therapy (Stage II-III, T2-4N0-3) or metastatic (M1; at least 80 pts).
5. At least one tumor lesion ≥ 10 mm.
6. At least one tumor lesion available for biopsy.
7. Newly diagnosed or confirmed progression and planned for therapy with trastuzumab emtansine or anti-HER2 targeted therapy(-ies) concomitant with chemotherapy (HER2-positive cohort) or chemotherapy (HER2-negative patients).
8. WHO performance status ≤ 2.
9. Predicted survival > 12 weeks.
10. Negative pregnancy test in women of childbearing potential (premenopausal or <12 months of amenorrhea post-menopause and who have not undergone surgical sterilization). Women of childbearing potential must use highly effective method of contraception, i.e combined hormonal contraception, or progestogen-only hormonal contraception, or intrauterine device, or intrauterine hormone-releasing system, or bilateral tubal occlusion, or vasectomized partner, or sexual abstinence

Exclusion Criteria:

1. Histologically or cytologically confirmed HER2-negative breast cancer defined as IHC 0 or 1+.
2. Other manifest malignancy.
3. Serious uncontrolled concomitant disease including congestive heart failure that would contraindicate the use of any anti-HER2 therapy.
4. Inadequate organ function, suggested by the following laboratory results:

   * Absolute neutrophil count <1,500 cells/mm3
   * Total bilirubin ≥1.5 x ULN (unless the patient has documented Gilbert's syndrome)
   * AST (SGOT) or ALT (SGPT) >5.0 × ULN
   * Serum creatinine clearance <30 ml/min
5. Patients of childbearing potential and sexually active and not willing to use highly effective contraceptive.
6. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
HER2- expression by using 68Ga-ABY-025 PET. | Approximately 10 days after study entry.
  HER2-expression in tumors measured by 68Ga-ABY-025 PET, centrally analysed and result used for location of biopsy.
HER2-expression by analysing biopsy sample. | Approximately 21 days after study entry.
  HER2-expression in tumors by histopathology. Location of biopsy site based on HER2 expression seen in ABY-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Lindman, Principal Investigator — Uppsala University Hospital
Locations (1):
- Section for Clinical Research & Development Unit, Uppsala, Sweden